CLINICAL TRIAL: NCT06336876
Title: Perceived Coping, Meaning, and Joy at Work
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 080.EDU.2019.R
Record Dates: First submitted 2020-09-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Undefined
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey Participant (Experimental): The sample will be a convenience sample of hospital-registered nurses and para-professional nursing services staff (e.g., patient care technicians and specialty area technicians) who agree to participate in an online survey launched via the Survey Monkey® portal.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Online survey launched via the Survey Monkey® portal

SUMMARY:
The aim of this study is to assess and describe employee characteristics associated with perceived horizontal inter-collegial workplace uncivil behavior within nursing services, and identify any relationships with meaning and joy in work (MJW), and assess job satisfaction.

DETAILED DESCRIPTION:
The study design is cross-sectional. This study will be conducted at a single Magnet-designated facility, Methodist Richardson Medical Center (MRMC), within the Methodist Health System. The sample will be a convenience sample of hospital-registered nurses and para-professional nursing services staff (e.g., patient care technicians and specialty area technicians) who agree to participate in an online survey launched via the Survey Monkey® portal. Survey Monkey® is an online, cloud-based survey delivery portal, and the subscription for the use of the portal is paid for by the Department of Education (DOE) at MRMC. Hence, the data will be owned by MHS. The study is a one-time inquiry. The PI and designated sub-investigators will send institutional emails to staff members who meet the inclusion criteria. The timeline for the study will be a total of four weeks. The study will be introduced for one week, be available for three weeks, and will conclude by the end of week four.

ELIGIBILITY:
Inclusion Criteria:

* The sample of participants will include all willing individuals who are registered nurses (full time, part time, and per-diem) Nursing para-professionals employed by Methodist Health System working at the MRMC campus and provide direct patient care for more than 50% of work hours
* All participants must be able to read and understand English.

Exclusion Criteria:

* employees who do not provide direct patient care for at least 50% of the time
* educators
* managers
* leaders
* advanced practice nurses
* non-nursing service personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Workplace Incivil Behavior | "through study completion, average of one year"
  [WIS, 7-item 4-point Likert scale with alpha, α 0.84 - 0.89]
Meaning, Joy in Work | "through study completion, average of one year"
  [MJW,17-item Likert scale with alpha,α 0.94]
Occupational Coping Self-Efficacy | "through study completion, average of one year"
  [OSCE-N, 9-item Likert scale with alpha, α- 0.83 to 0.97]
Demographic | "through study completion, average of one year"
  10-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Adegbola, RN, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No